CLINICAL TRIAL: NCT07068854
Title: New Insights Into the Development and Biological Activity Evaluation of Mango Juices Processed by Sustainable Emerging Technologies
Brief Title: New Insights Into the Biological Activity Evaluation of Mango Juices Processed by Sustainable Emerging Technologies
Acronym: BIOACTIMANGO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Concepción Sánchez-Moreno, Dr., National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PID2023-147025NB-I00
Record Dates: First submitted 2025-06-24; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Biomarkers of Food Intake in Healthy Subjects
Keywords: Mango juice; Phytochemicals; Bioavailability; Biomarkers; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPP mango juice (Experimental): mango puree (20%)-orange juice (80%)
  Interventions: Other: HPP mango juice group
- control juice (Experimental): water (20%)-HPP orange juice (80%)
  Interventions: Other: control juice

INTERVENTIONS:
Other: HPP mango juice group — During each intervention period, participants will be instructed to consume 500 mL of juice/day in two doses, 250 mL in the morning and 250 mL in the afternoon
  Arms: HPP mango juice
Other: control juice — During each intervention period, participants will be instructed to consume 500 mL of juice/day in two doses, 250 mL in the morning and 250 mL in the afternoon
  Arms: control juice

SUMMARY:
The aim of this clinical trial is to study the effect of a habitual dietary intake of commercial high pressure-processed (HPP) mango juice [mango puree (20%)-orange juice (80%)] or control juice [water (20%)-HPP orange juice (80%)]. There are numerous in vitro and in vivo animal studies that support exceptional health-promoting characteristics of mango products (pulp, peel, seed, juice, extracts, etc.) such as antidiabetic, anticancer, antiinflammatory, antioxidant and antibacterial activities based on their phytochemical composition, but there are many fewer studies assessing the absorption, metabolism, and health-related properties of phytochemical from commercial mango fruit juices (only 20% of mango pulp) in humans. Consequently, this study proposes for the first time the study of the effects of commercial HPP mango juice consumption on health biomarkers by a human intervention study. Researchers will compare the bioavailability (metabolite profiles) of compounds with health effects and the biomarkers of health to evaluate if mango juice works better that control juice.

DETAILED DESCRIPTION:
The human intervention study has been designed with the aim to study the effect of a usual dietary intake of a commercial HPP mango juice on phenolic and carotenoid compounds bioavailability and health-related biomarkers. Due to mango juice is obtained from a pulp puree, the high viscosity of this product makes it necessary to mix it with water or other fruit juice for consumption. Thus, the commercial mango juice is not actually composed of 100% mango. For the present study, it has been selected a commercial HPP mango juice whose composition is mango puree 20% and orange juice 80%. A commercial HPP orange juice 100% elaborated with the same process will be consumed by the participants as control juice after be diluted. Subjects will be instructed to dilute the commercial HPP orange juice with water to match the content of orange juice in both groups. A 28-day feeding trial (randomized cross-over controlled clinical trial) will be conducted to study the effect of a usual dietary intake of commercial HPP mango juice [mango puree (20%)-orange juice (80%)] or control juice [water (20%)-HPP orange juice (80%)] on phenolic and carotenoid metabolite profiles and cardiometabolic health biomarkers. To date, no human intervention studies have been conducted to assess the health effects of ingesting commercial HPP-treated mango juices.

Recruitment of study participants. The inclusion criteria will be: individuals with body mass index [BMI] 25-29.9, aged 18-50, plasma total cholesterol levels 180-235 mg/dL, and plasma retinol concentration in the upper tertile of the normal reference range (20-60 µg/dL). Subjects will be recruited at the Human Nutrition Unit (HNU), Institute of Food Science, Technology and Nutrition (ICTAN). The study will be advertised at the campus of Universidad Complutense de Madrid (UCM), on the webpage of ICTAN-CSIC and through different social media. All participants will attend a familiarization session before beginning the study. The exclusion criteria will be: use of medication/food supplements to lower blood cholesterol, chronic disease, such as high blood pressure, diabetes, and heart disease; pregnancy or lactation; smoking habits; alcohol consumption above recommendations; allergy to mango or orange fruit.

Study design and dietary intervention. The participants will receive oral and written information about the study and provide written consent. This study will be a randomized cross-over controlled clinical trial. Approval by the Ethics Committee for Clinical Research of the University Hospital Puerta de Hierro Majadahonda, Spain has been obtained. To avoid sex and gender bias, men and women will be recruited. Subjects will be randomly to either the HPP mango juice group or the control juice group. Each intervention period will last 4 weeks and will be separated by a 4-week wash-out period. During each intervention period, participants will be instructed to consume 500 mL of juice/day in two doses, 250 mL in the morning and 250 mL in the afternoon. Daily dose of juice (500 mL) and duration of intervention (4 weeks) have been selected based on our previous human intervention studies and literature studies, both compatible with a usual dietary intake. Three visits to HNU at ICTAN will be required by the study protocol: the initial screening, at Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28). Participants will be fasted overnight. On study visit days to HNU at ICTAN, fasting blood samples will be drawn, urine and faeces samples will be collected. It is planned that a total of 30 individuals will be recruited to obtain outcome significant differences. The primary outcome variable for sample size calculation has been the modification in the plasma CRP levels (as inflammation biomarker). In particular, power calculations have been based on a 30% reduction in CRP levels following previous nutritional clinical trials in subjects consuming fruit juices containing mango, orange or similar. A sample size of 30 has been calculated as sufficient to detect this change with 95% power and an alpha value of 0.05, using published variances of this parameter. Blood samples will be drawn and collected on days 0, 14, and 28 of the study. Urine and faeces will be collected the same days of blood sample collection and stored at -80 °C until analysis.

The following determinations will be performed at different periods: anthropometric measurements and blood pressure, dietary analysis; phenolic and carotenoid compounds analysis in plasma/serum/urine, carotenoid compounds analysis in serum and faeces, lipid profile and biochemistry markers, inflammatory and vascular injury biomarkers and metabolic hormones, oxidative stress biomarkers, and antioxidant enzyme activities and plasma antioxidant activity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [BMI] 25-29.9 kg/m^2
* Age 18-50 years
* Plasma total cholesterol levels 180-235 mg/dL
* Plasma retinol concentration in the upper tertile of the normal reference range (20-60 µg/dL)

Exclusion Criteria:

* Use of medication/food supplements to lower blood cholesterol
* Chronic disease, such as high blood pressure, diabetes, and heart disease
* Pregnancy or lactation
* Smoking habits
* Alcohol consumption above recommendations
* Allergy to mango or orange fruit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein (CRP) | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma CRP levels as result of HPP mango juice intake

SECONDARY OUTCOMES:
BMI | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of BMI as result of HPP mango juice intake
Body weight | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of body as result of HPP mango juice intake
Pulse | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of pulse as result of HPP mango juice intake
Temperature | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of temperature as result of HPP mango juice intake
Systolic blood pressure | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of systolic blood pressure as result of HPP mango juice intake
Diastolic blood pressure | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of diastolic blood pressure as result of HPP mango juice intake
Phenolic and carotenoid compounds | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of blood and urinary/faecal phenolic and carotenoid metabolites as result of HPP mango juice intake
Total cholesterol | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma total cholesterol as result of HPP mango juice intake
HDL-cholesterol | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma HDL-cholesterol as result of HPP mango juice intake
LDL-cholesterol | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma LDL-cholesterol as result of HPP mango juice intake
VLDL-cholesterol | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma VLDL-cholesterol as result of HPP mango juice intake
Triacylglycerols | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma triacylglycerols as result of HPP mango juice intake
Glucose | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma glucose as result of HPP mango juice intake
Urea | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma urea as result of HPP mango juice intake
Uric acid | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma uric acid as result of HPP mango juice intake
Creatinine | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma creatinine as result of HPP mango juice intake
Albumin | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma albumin as result of HPP mango juice intake
Alanine aminotransferase (ALT/GPT) | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma alanine aminotransferase (ALT/GPT) as result of HPP mango juice intake
Aspartate aminotransferase (AST/GOT) | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma aspartate aminotransferase (AST/GOT) as result of HPP mango juice intake
Gamma-glutamyl transpeptidase (GGT) | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma gamma-glutamyl transpeptidase (GGT) as result of HPP mango juice intake
Total bilirubin | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma total bilirubin as result of HPP mango juice intake
Inflammatory and vascular injury biomarkers and metabolic hormones | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma inflammatory cytokines, cardiovascular biomarkers and metabolic hormones as result of HPP mango juice intake
Oxidative stress biomarkers | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of plasma oxidative stress biomarkers as result of HPP mango juice intake
Antioxidant enzyme activities and antioxidant activity | At Week 0 (day 0-Baseline), and Weeks 2 (day 14), and 4 (day 28)
  Changes of erythrocyte superoxide dismutase (SOD), catalase (CAT) and glutathione peroxidase (GPx) activities as result of HPP mango juice intake. Changes of plasma 2,2'-azinobis(3-ethylbenzothiazoline-6-sulfonic acid) radical cation (ABTS•+) scavenging capacity and ferric reducing antioxidant power (FRAP) as result of HPP mango juice intake
Dietary analysis | At Week 0 (day 0-Baseline) of each of the two intervention periods
  Participants will be asked to maintain their dietary habits, except for the daily mango and orange supplementation. The overall dietary intake of each subject will be evaluated using three 24-h diet recall (two weekdays and one weekend day) at the beginning of each of the two intervention periods to analyse the intakes of total energy, carbohydrate, protein, and fat; and total phenolic compounds and total carotenoid compounds

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food Science, Technology and Nutrition (ICTAN), National Research Council (CSIC), Madrid, Madrid, Spain